CLINICAL TRIAL: NCT00574210
Title: A Randomized, Double-blind, Placebo-controlled, 5-arm Parallel Study to Evaluate the Pharmacokinetics/ Pharmacodynamics and Steady State Efficacy of Once or Twice Daily Bilastine (10 or 20 mg) Compared With Placebo Given Orally in the Treatment of the Symptoms of Seasonal Allergic Rhinitis in an Environmental Exposure Chamber (EEC) Mode
Brief Title: PK/PD and Steady State Efficacy Study of Bilastine Compared With Placebo Given Orally in the Treatment of the Symptoms of SAR in an EEC Model (5-arm)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: Allied Research International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 2507/EEC; P2FZ07001
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Allergic Rhinitis; Hay Fever; Rhinoconjunctivitis
Keywords: Seasonal Allergic Rhinitis (SAR); Environmental Exposure Chamber (EEC); Therapeutic Uses; Antihistamine Drug; Ragweed Pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — bilastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Bilastine oral 20 mg once per day (1 x 20 mg bilastine tablet plus 1 placebo tablet)
  Interventions: Drug: Bilastine
- 2 (Experimental): Bilastine oral 20 mg twice per day (2 x 20 mg bilastine tablets)
  Interventions: Drug: Bilastine
- 3 (Experimental): Bilastine oral 10 mg once per day (1 x 10 mg bilastine tablet plus 1 placebo tablet)
  Interventions: Drug: Bilastine
- 4 (Experimental): Bilastine oral 10 mg twice per day (2 x 10 mg bilastine tablets)
  Interventions: Drug: Bilastine
- 5 (Placebo Comparator): Placebo oral twice per day (2 placebo tablets)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Bilastine Tablets, administered at a dosage strength of 10 mg or 20 mg, once or twice per day.
  Arms: 1; 2; 3; 4
Drug: Placebo — Placebo Tablets administered twice per day
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the relative efficacy of four dosing regimens of bilastine tablets versus placebo in subjects with SAR exposed in controlled ragweed pollen using the EEC model based on the mean change from baseline in Total Nasal Symptom Scores (TNSS). Study includes male and female subjects, aged 18 and 65 years with clinical history of SAR with seasonal onset and offset of nasal allergy symptoms during each of the last two ragweed allergy seasons and a positive skin prick test to ragweed allergen within 12 months prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of SAR for the last two ragweed allergy seasons.
* A positive skin test within 12 months of screening to ragweed allergen.
* A minimum qualifying symptom score on both Visits, 2 and 3.
* Females must have a confirmed absence of pregnancy according to a negative urine pregnancy test.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning a pregnancy.
* History of more than mild asthma.
* History of clinically significant (as determined by the Investigator) active perennial allergic rhinitis to which the subject is regularly exposed.
* Non-allergic rhinitis (vasomotor or rhinitis medicamentosa).
* An anatomic abnormality that interferes with assessment of nasal function. - History of clinically significant recurrent sinusitis or chronic sinusitis. - Clinically significant (as determined by the Investigator) cardiovascular, hepatic, neurologic, psychiatric, endocrine, or other significant systemic disease that makes implementation of the protocol jeopardizing to the safety of the subject.
* A need for use of antihistamines or corticosteroids on a regular basis (systemic or topical).
* Currently taking monoamine oxidase (MAO) inhibitors.
* Taken any systemic corticosteroids, immunomodulators, or immune suppressive medications within four weeks prior to Visit 1.
* Taken any antihistamine within seven days prior to Visit 1 skin testing.
* Known current alcohol or drug abuse.
* Current participation in another clinical study involving an experimental treatment, or participation in such a study within 30 days prior to study entry. - History of generalized anaphylaxis requiring medical attention.
* Clinically significant abnormality of screening blood chemistry, hematology, or urinalysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Scores (TNSS) | within 10 days

SECONDARY OUTCOMES:
Total Symptom Scores (TSS), Total Non-Nasal Symptom Scores (TNNSS), Total Ocular Symptoms Scores (TOSS), Area Under the Curve (AUC) of TNSS, TSS, TOSS, TNNSS, Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ - EEC) | witin 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Roman Valiente, MD, Study Chair — Faes Farma, S.A.; Piyush Patel, MD, Study Director — Allied Research International Inc; Deepen Patel, MD, CCFP, Principal Investigator — Allied Research International Inc
Locations (1):
- Allied Research International - Cetero Research, Mississauga, Ontario, Canada